CLINICAL TRIAL: NCT01863030
Title: A Prospective, Observational Study Utilizing Phasix™ Mesh During Ventral and Incisional Hernia Repair Surgery
Status: Completed | Type: Observational
Sponsor: John Roth (Other)
Responsible Party: Sponsor-Investigator, John Roth, PI, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: Phasix
Record Dates: First submitted 2013-05-14; First posted 2013-05-27 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Ventral Hernia
Keywords: Resorbable mesh; Phasix mesh
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Phasix mesh: Mesh being used for approved use. Mesh for ventral and incisional hernias.
  Interventions: Device: Phasix mesh implant

INTERVENTIONS:
Device: Phasix mesh implant

SUMMARY:
The objective of this study is to collect efficacy, safety and utility data with Phasix™ Mesh in ventral and incisional repair procedures by evaluating the following:

1. Hernia recurrence rate of ventral and incisional hernias post repair with Phasix™ Mesh for up to 12 months post surgery.
2. Perioperative, short-term and long-term procedural and/or device related complications.
3. Abdominal Wall Function and mobility.

ELIGIBILITY:
Inclusion Criteria:

The subject must meet all of the relevant criteria listed below to be enrolled in the study:

1. Subject must be ≥18 years of age.
2. Subject or subject's legally authorized representative must be willing give written informed consent.
3. Subject must be diagnosed with a ventral, incisional or first-recurrent incisional hernia.
4. Hernia size greater than 10cm2 and less than 250cm2
5. Subject must be willing to undergo ventral hernia repair and be able to undergo all other study procedures as outlined in this protocol.

Exclusion Criteria:

The subject must be excluded from study enrollment if any of the following criteria are met:

1. Subject's hernia is multiply recurrent.
2. CDC wound classification other than clean or clean-contaminated
3. The use of surgical repair as a bridge.
4. Patient has a contraindication to placement of mesh.
5. Concomitant procedures with wound classification other than clean
6. Subject has peritonitis.
7. Subject is on or suspected to be placed on chemotherapy medications during any part of the study.
8. Subject's body mass index (BMI) >55 kg/m2.
9. Subject has cirrhosis, and/or ascites.
10. Subject is American Society of Anesthesiology Class 4 or 5.
11. Subject is known to be infected with human immunodeficiency virus (HIV).
12. Subject has known allergies to tetracycline or kanamycin.
13. Subject has a life expectancy of less than 2 years at the time of enrollment.
14. Subject has any condition in the opinion of the Investigator that would preclude the use of the study device, or preclude the subject from completing the follow-up requirements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patents with ventral hernias that meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John S Roth, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plymale MA, Davenport DL, Dugan A, Zachem A, Roth JS. Ventral hernia repair with poly-4-hydroxybutyrate mesh. Surg Endosc. 2018 Apr;32(4):1689-1694. doi: 10.1007/s00464-017-5848-7. Epub 2017 Sep 15. PMID 28916979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with a diagnosis of a ventral or incisional hernia requiring surgical repair to close the defect were recruited. First subject enrolled June 2013. The last subject was enrolled August 2014.
Groups:
- Phasix Mesh: Phasix mesh implant
Period: Baseline
Arm/Group | Phasix Mesh
Started | 31
Completed | 31
Not Completed | 0
Period: Follow up
Arm/Group | Phasix Mesh
Started | 31
2 Weeks | 31
3 Months | 28
6 Months | 29
12 Months | 26
24 Months | 13
Completed | 13
Not Completed | 18

BASELINE CHARACTERISTICS:
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 52 [44 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 28
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 33 [28.6 to 38.4]
Employment Status [Count of Participants; unit: Participants]
  Employed | 12
  Unemployed/retired | 11
  Disabled | 8
Employment Activity [Count of Participants; unit: Participants]
  Manual Labor | 6
  Sedentary | 5
  not employed | 19
  Employment activity not answered | 1
Past Medical History [Count of Participants; unit: Participants]
  Cancer | 5
  Peripheral Vascular Disease | 1
  Chronic Heart Failure/ Coronary Artery Disease | 5
  GERD | 12
  COPD | 9
  Diabetes | 8
  Genitourinary disease | 5
  Mental Health Disease | 4
  Chronic Pain | 10
Number of Participants with History of Tobacco Use [Count of Participants; unit: Participants] | 7
Prior Abdominal Surgery [Count of Participants; unit: Participants] | 30
Prior Hernia Repair [Count of Participants; unit: Participants] | 14
Operation Duration [Median (Inter-Quartile Range); unit: Minutes] | 140 [118 to 179]
CDC Wound Classification [Count of Participants; unit: Participants] — CDC wound class Class 1: An uninfected operative wound in which no inflammation is encountered. Class 2: An operative wound in which the respiratory, alimentary, genital, or urinary tracts are entered under controlled conditions and without unusual contamination. Class 3: Open, fresh, accidental wounds. Operations with major breaks in sterile technique or gross spillage from the gastrointestinal tract. Incisions with acute, nonpurulent inflammation. Class 4: Old traumatic wounds with retained devitalized tissue. Those that involve existing clinical infection or perforated viscera.
  Participants
    Grade 1 | 30
    Grade 2 | 1
Removal of Previous mesh during hernia repair procedure [Count of Participants; unit: Participants] — Removal of previous mesh that was in place prior to enrollment.
  Participants | 4
Hernia Defect Size [Median (Inter-Quartile Range); unit: cm2] — Size of the hernia defect before repair. Measured during hernia repair procedure.
  cm2 | 105 [74 to 130]
Graft Size [Median (Inter-Quartile Range); unit: cm2] | 592 [388 to 643]
Number of Grafts used [Count of Participants; unit: Participants]
  1 graft | 30
  2 grafts | 1
Number of Participants with Retro Rectus Mesh Placement [Count of Participants; unit: Participants] — Number of participants in which the mesh is placed above the posteriorrectus sheath and below the muscle.
  Participants | 31
Component Separation Technique [Number; unit: participants]
  Open CST | 31
  Endo CST | 30
  Posterior CST | 18
  Rives Stoppa | 11
Number of Participants with Posterior Rectus Sheath Approximation [Count of Participants; unit: Participants] — Number of participants in which the two sides of the posterior sheaths are sewn together in entirety.
  Participants | 31
Number of Participants with Anterior Rectus Sheath Approximation [Count of Participants; unit: Participants] — Number of participants in which both the right and left side of the sheath are sewn together with no gaps.
  Participants | 31
Number of participants where PDS sutures were used during hernia repair procedure [Count of Participants; unit: Participants] | 31
Number of participants who had drains placed during hernia repair procedure [Number; unit: participants]
  1 drain | 10
  2 drains | 19
  3 drains | 2
Number of participants who had a concurrent procedure [Count of Participants; unit: Participants] — Number of participants who had a concurrent procedure at the same time as the index hernia repair procedure.
  Participants | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrent Ventral and Incision Hernias Post Repair With Phasix™ Mesh
Description: Number of participants with recurrent ventral and incision hernias post repair with Phasix™ Mesh. Hernia recurrence is measured by physical exam.
Time Frame: up to 24 months post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
Participants | 0

2. Other Pre Specified Outcome: Physical Component Summery
Description: Quality of life survey- Short Form 12. Physical component summery. Assessment of physical limitations such as bathing, dressing, or physical activities. Scales range from 0-100. Low scores indicate someone with many limitations, while high scores indicate someone with no or few limitations.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 38.9 (10.0)
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 47.2 (9.7)
  24 months post operation: number analyzed (Participants) | 15
  24 months post operation | 43.9 (9.4)

3. Other Pre Specified Outcome: Role Emotional Quality of Life Outcome
Description: Quality of life survey- Short Form 12 Role emotional subdomain. This assesses if the patient experiences problems with work or other daily activities as a result of their emotional health. Scales range from 0-100. Low scores indicate the patient experiences many problems at work or with other daily activities as a result of poor emotional health. High scores indicate no problems with work or daily activities as a result of emotional health.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 42.5 (12.9)
  12 months post operation | 43.5 (13.0)
  24 months post operation | 44.8 (12.0)

4. Other Pre Specified Outcome: Physical Functioning Quality of Life Outcome
Description: Quality of life survey- Short Form 12 Physical Functioning subdomain. Assesses ability to perform physical activities, including bathing and dressing one's self. Scales range from 0-100. Low scores indicate many limitations with physical activities. High scores indicate no problems with physical activities.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 39.8 (12.1)
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 46.4 (11.6)
  24 months post operation: number analyzed (Participants) | 15
  24 months post operation | 44.5 (12.2)

5. Other Pre Specified Outcome: Role Physical Quality of Life Outcome
Description: Quality of life survey- Short Form 12 Role physical subdomain. Assesses ability to perform physical activity such as bathing and dressing one's self. Scales range from 0-100. Low scores indicate problems with physical activities. High scores indicate no problems performing physical activities.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 39.0 (11.7)
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 46.1 (44.2)
  24 months post operation: number analyzed (Participants) | 15
  24 months post operation | 44.2 (11.1)

6. Other Pre Specified Outcome: Bodily Pain Quality of Life Outcome
Description: Quality of life survey- Short Form 12 Bodily Pain subdomain. Assesses level of bodily pain. scales range from 0-100. low scores indicate a severe level of pain that is limiting. High scores indicate a low level of pain or no pain-related limitations.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 38.5 (12.7)
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 45.9 (11.1)
  24 months post operation: number analyzed (Participants) | 15
  24 months post operation | 44.5 (13.1)

7. Other Pre Specified Outcome: General Health Quality of Life Outcome
Description: Quality of life survey- Short Form 12 General Health Subdomain. Assesses level of general health related to . Scales 0-100. low scores indicate poor general health, and high scores indicate good general health.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 43.3 (91)
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 50.7 (10.4)
  24 months post operation: number analyzed (Participants) | 15
  24 months post operation | 43.9 (12.6)

8. Other Pre Specified Outcome: Mental Component Summery
Description: Quality of life survey- Short Form 12 Mental Component Summery. Assesses level of mental health. Scales range from 0-100. Low scores indicate nervousness and depression. High scores indicate feeling peaceful, happy, and calm.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 46.5 (11.7)
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 48.3 (9.8)
  24 months post operation: number analyzed (Participants) | 15
  24 months post operation | 47.9 (10.9)

9. Other Pre Specified Outcome: Vitality Quality of Life Outcome
Description: Quality of life survey- Short Form 12 Vitality subdomain. Assesses level of energy. Scales range from 0-100. Low scores indicate low levels of energy, while high scores indicate high levels of energy.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 45.3 (12.1)
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 50.2 (9.8)
  24 months post operation: number analyzed (Participants) | 15
  24 months post operation | 47.1 (10.0)

10. Other Pre Specified Outcome: Social Functioning Quality of Life Outcome
Description: Quality of life survey- Short Form 12 Social Functioning subdomain. Assesses ability to participate in normal social activities without difficulties due to physical or emotional health problems. Scores are normalized to 0-100, with 50 being the national normalized mean. Lower scores indicate many difficulties with normal social activities due to physical or emotional health problems. Higher scores indicate little or no difficulties with normal social activities due to physical or emotional health problems.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 43.4 (12.1)
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 47.0 (11.3)
  24 months post operation: number analyzed (Participants) | 15
  24 months post operation | 48.6 (9.8)

11. Other Pre Specified Outcome: Mental Health Quality of Life Outcome
Description: Quality of life survey- Short Form 12 Mental Health subdomain. assesses level of mental health. Scale ranges from 0-100. Low scores indicate depression and nervousness. High scores indicate feeling peaceful, happy, and calm.
Time Frame: baseline, 12 months, 24 months
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 12 months and 24 months post operation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  Baseline/ pre operation | 45.3 (13.3)
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 50.3 (8.5)
  24 months post operation: number analyzed (Participants) | 15
  24 months post operation | 47.0 (14.2)

12. Other Pre Specified Outcome: Abdominal Wall Mobility
Description: Abdominal wall strength will be measured using the trunk mobility measurements, curl up performance test and EPIC lift capacity test preoperatively, 3 months (+/- 1 month) postoperatively and 12 months postoperatively.
Time Frame: 12 Months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Abdominal Wall Function
Description: as for outcome 12
Time Frame: up to 12 months post surger
Reporting Status: Not Posted

14. Post Hoc Outcome: Pain Assessment
Description: Pain rating on a numeric rating scale (0=no pain, 10=extreme pain)
Time Frame: up to 24 months post surgery
Population: 31 patients were implanted with phasix mesh. Patients were lost to follow up at 3 months, 6 months, 12 months, and 24 months post operation.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  2 weeks post operation | 4.0 [2.0 to 6.0]
  3 months post operation: number analyzed (Participants) | 28
  3 months post operation | 1.0 [1.0 to 4.0]
  6 months post operation: number analyzed (Participants) | 29
  6 months post operation | 1.0 [1.0 to 2.0]
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 1.0 [1.0 to 3.8]
  24 months post operation: number analyzed (Participants) | 13
  24 months post operation | 2.5 [1.0 to 5.5]

15. Post Hoc Outcome: Tenderness Assessment
Description: Tenderness measure on a numeric rating scale (0=no tenderness, 10= extreme tenderness)
Time Frame: 24 months
Population: 31 patients were implanted. patients were lost to follow up at 3 months, 6 months, 12 months, and 24 months post operation.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Phasix Mesh
Number analyzed (Participants) | 31
units on a scale
  2 weeks post operation | 3.0 [1.0 to 4.0]
  3 months post operation: number analyzed (Participants) | 28
  3 months post operation | 1.0 [1.0 to 2.0]
  6 months post operation: number analyzed (Participants) | 29
  6 months post operation | 1.0 [1.0 to 3.0]
  12 months post operation: number analyzed (Participants) | 26
  12 months post operation | 1.0 [1.0 to 1.0]
  24 months post operation | 1.0 [1.0 to 1.0]

ADVERSE EVENTS:
Time Frame: 3 years, 3 months, 9 days
Arm/Group | Phasix Mesh
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 6/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phasix Mesh (N=31)
Seroma (Surgical and medical procedures) | 4 (4)
Wound Dehiscence (Surgical and medical procedures) | 1 (1)
Soft Tissue Necrosis (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No